CLINICAL TRIAL: NCT07279753
Title: Effects of a Critical Thinking-Based Tactical Training Program on Tactical Skills and Futsal-Specific Performance in University Players: A Single-Group Pre-Post Study
Brief Title: Critical Thinking Tactical Training in University Futsal Players
Acronym: TPCT-FUTSAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Responsible Party: Principal Investigator, Édison Andrés Pérez Bedoya, Principal Investigator, Lecturer in Physical Education, Federal University of Vicosa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TdeA-USBMed-TPCT-FUTSAL
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Athletic Performance; Decision Making
Keywords: Futsal; Tactical Training; Critical Thinking; Team Sports; University Athletes; Performance Analysis

STUDY DESIGN:
Intervention Model Description: Single-group, pre-post interventional model. A single cohort of university futsal players receives the critical thinking-based tactical training program, with all participants exposed to the same sequence of training sessions. Tactical and performance outcomes are assessed before and after the intervention, and each participant serves as his own control. No randomization or parallel comparison group is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPCT (Experimental): This arm includes a single cohort of university futsal players who receive a critical thinking-based tactical training program (TPCT). The intervention is delivered during regular team training over multiple weeks through structured sessions that combine dynamic warm-up, representative small-sided games, and futsal-specific tactical scenarios. Each session uses guided discovery and reflective questioning to promote tactical awareness, anticipation, and collective decision-making. Task constraints, game formats, and intensity are progressively adjusted to increase tactical complexity and physiological load during the main training blocks. All enrolled participants receive the same intervention, and each player serves as his own control through pre- and post-intervention assessments.
  Interventions: Other: Tactical Program Critical Thinking

INTERVENTIONS:
Other: Tactical Program Critical Thinking — The intervention is a futsal-specific tactical training program structured around critical thinking (TPCT). Across multiple weeks, players complete representative small-sided and conditioned games framed by brief tactical problems (for example, creating numerical superiority or protecting central lanes). During tasks, the coach uses guided discovery and structured questioning to promote reading of key cues, generation and comparison of options, justification of decisions using principles of play, and anticipation of opponents' and teammates' actions. Task constraints and intensity are progressively adjusted, and each session ends with a brief collective reflection.

SUMMARY:
This study examined the effects of a tactical training program based on critical thinking (TPCT) on the tactical efficiency and decision-making performance of university futsal players. The intervention was designed to strengthen players' ability to interpret the dynamics of play, anticipate opponents' actions, and generate adaptive tactical responses under competitive conditions.

The program followed a socio-constructivist framework, promoting learning through problem solving and interaction among teammates. Training sessions combined representative game situations, reflective questioning, and guided tactical discussions.

A single-group pre-post design was implemented. Thirteen university players participated voluntarily after providing informed consent and receiving approval from the institutional ethics committee. Data were collected before and after the intervention to assess individual and collective tactical performance, goal effectiveness, and time of ball possession.

The study aimed to provide evidence on the educational and performance impact of a critical thinking-based tactical approach in futsal, contributing to contemporary models of athlete development and pedagogical innovation in team sports.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of enrollment.
* Registered player of the university futsal team participating in the study.
* Minimum of 1 year of regular, organized futsal practice.
* Regular attendance at team training (at least 2 sessions per week) in the 3 months prior to baseline testing.
* Medical clearance or self-report indicating ability to perform high-intensity futsal training and testing.
* Provision of written informed consent.

Exclusion Criteria:

* Current musculoskeletal injury or pain that limits normal futsal training or match participation at baseline.
* History or diagnosis of cardiovascular, respiratory, neurological, or metabolic disease that contraindicates high-intensity exercise.
* Use of medications that substantially affect physical performance, heart rate response, or perception of effort, as judged by the study physician or medical screener.
* Participation in another structured experimental training program targeting futsal performance during the intervention period.
* Absence from more than 20% of the scheduled TPCT training sessions.
* Withdrawal of informed consent at any time during the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participation is not restricted based on self-identified gender. Eligibility is defined by biological sex and membership in the university futsal team according to the study inclusion criteria, without additional limitations based on gender identity.
Enrollment: 13 (Actual)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Change in execution time during futsal-specific tactical test | Time Frame: Baseline (up to 7 days before the first TPCT session) and post-intervention (up to 7 days after the final TPCT session), up to 7 weeks in total
  Time (seconds) required for each player to complete a standardized futsal-specific tactical test involving ball control, passing, movement, and finishing actions in a predefined sequence. The test is administered individually under stable conditions. The primary endpoint is the change in execution time from pre- to post-intervention; lower times indicate better tactical-motor efficiency and faster resolution of the game situation.

SECONDARY OUTCOMES:
Change in number of goals scored during futsal-specific tactical test | Time Frame: Baseline (up to 7 days before the first TPCT session) and post-intervention (up to 7 days after the final TPCT session), up to 7 weeks in total
  Number of goals scored by each player during a standardized futsal-specific tactical test, performed under the same conditions at baseline and post-intervention. The test requires completing a predefined sequence of actions (ball control, passing and finishing) with a fixed number of shooting opportunities. The secondary endpoint is the change in goals scored from pre- to post-intervention; higher values indicate better offensive effectiveness during the test.
Change in the quality of collective tactical discourse during TPCT sessions | Time Frame: Week 2 and Week 7 of the TPCT programme (early and late intervention sessions; approximately 6-7 weeks)
  Change in the quality of collective tactical discourse during TPCT sessions, analysed from two audio-recorded group discussions (early and late intervention). Transcripts are segmented into turns of talk or thematic fragments and coded with a 10-indicator analytic rubric (0-3 scale) derived from the TPCT (e.g., clarity of objective, contextual specificity, anticipation, counter-argumentation, integration of perspectives, metacognition). Session-level scores and deltas (late-early) are computed, and emergent themes (for example time management, responsibility, commitment) are described to complement quantitative performance outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de San Buenaventura - Medellín, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not been finalized. The study involves a small, identifiable sample of university athletes from a single team, which increases the risk of re-identification even after de-identification procedures. Before any IPD can be shared, the research team must review the informed consent documentation, institutional policies, and ethics committee recommendations to determine whether controlled access to an anonymized dataset is appropriate. If IPD sharing is implemented in the future, conditions for access, type of data shared, and repository details will be specified in an updated record and in subsequent publications.